CLINICAL TRIAL: NCT00588861
Title: Total Hip Replacement With the Answer® Hip Stem and Ranawat/Burnstein® Acetabular Shell Using Simplex® or Palacos® Bone Cement
Brief Title: Total Hip Replacement With the Answer® Hip Stem and Ranawat/Burnstein® Shell Using Simplex® or Palacos® Bone Cement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to insufficient data and lack of patient follow-up
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-U-011
Record Dates: First submitted 2007-12-19; First posted 2008-01-09 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis, Hip; Traumatic Arthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Answer® hip stem with Simplex Cement (Active Comparator): Femoral stem replacement with Answer® hip stem & Simplex Bone Cement
  Interventions: Device: Answer® hip stem
- Answer® hip stem with Palacos Cement (Active Comparator): Femoral stem replacement with Answer® hip stem & Palacos Bone Cement
  Interventions: Device: Answer® hip stem

INTERVENTIONS:
Device: Answer® hip stem — Total hip replacement using Palacos® bone cement, the Answer® hip stem and the Ranawat/Burnstein® acetabular shell.
  Other Names: Answer Hip Stem; Simplex Bone Cement
Device: Answer® hip stem — Total hip replacement using Simplex® bone cement, the Answer® hip stem and the Ranawat/Burnstein® acetabular shell.
  Other Names: Answer Hip Stem; Palacos Bone Cement

SUMMARY:
The purpose of this study is to document the clinical outcomes of several devices used in total hip replacement, including the Answer® hip stem, the Ranawat/Burnstein® acetabular shell, and Simplex® or Palacos® bone cement.

DETAILED DESCRIPTION:
The purpose of this study is to document the clinical outcomes of several devices used in total hip replacement, including the Answer® hip stem, the Ranawat/Burnstein® acetabular shell, and Simplex® or Palacos® bone cement. It was desirable to see if there were any differences in the outcomes of two different types of bone cement in application.

ELIGIBILITY:
Inclusion Criteria:

* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable using other techniques

Exclusion Criteria:

* Infection, sepsis, and osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Beres, MD, Study Director — Zimmer Biomet
Locations (1):
- Biomet Orthopedics, LLC, Warsaw, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by the investigator based on the FDA cleared inclusion/exclusion criteria in the protocol.
Pre-assignment Details: The patients were assigned to each group according to the bone cement used with the implant.
Groups:
- Answer Stem Utilizing Simplex Cement: Simplex Cement is a bone cement used for implant fixation. It is a powder premixed with antibiotics
- Answer Stem Utilizing Palacos Cement: Palacos Cement is bone cement used to secure artificial implants to bone that has a green color in order to improve visualization during implantation.
Period: Pre-Operative
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 202 (202 Patients were enrolled, however only 107 contributed preop data.) | 200 (200 patients were enrolled, however only 114 contributed preop data.)
Completed | 107 | 114
Not Completed | 95 | 86
Not completed — Patients Did Not Complete Preop Data | 95 | 86
Period: 6 Months
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 6 Months, however only 9 returned for follow-up.) | 114 (114 cases were due at 6 Months, however only 41 returned for follow-up.)
Completed | 9 | 41
Not Completed | 98 | 73
Not completed — Patients did not return for follow-up | 98 | 73
Period: 1 Year
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 1 Year, however only 18 returned for follow-up.) | 114 (114 cases were due at 1 Year, however only 32 returned for follow-up.)
Completed | 18 | 32
Not Completed | 89 | 82
Not completed — Patients did not return for follow-up | 89 | 82
Period: 2 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 2 Years, however only 15 returned for follow-up.) | 114 (114 cases were due at 2 Years, however only 27 returned for follow-up.)
Completed | 15 | 27
Not Completed | 92 | 87
Not completed — Patients did not return for follow-up | 92 | 87
Period: 4 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 4 Years, however only 16 returned for follow-up.) | 114 (114 cases were due at 4 Years, however only 11 returned for follow-up.)
Completed | 16 | 11
Not Completed | 91 | 103
Not completed — Patients did not return for follow-up | 91 | 103
Period: 6 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 6 Years, however only 3 returned for follow-up.) | 114 (114 cases were due at 6 Years, however only 5 returned for follow-up.)
Completed | 3 | 5
Not Completed | 104 | 109
Not completed — Patients did not return for follow-up | 104 | 109
Period: 8 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 8 Years, however only 2 returned for follow-up.) | 114 (114 cases were due at 8 Years, however no patients returned for follow-up.)
Completed | 2 | 0
Not Completed | 105 | 114
Not completed — Patients did not return for follow-up | 105 | 114
Period: 10 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Started | 107 (107 cases were due at 10 Years, however no patients returned for follow-up.) | 114 (114 cases were due at 10 Years, however no patients returned for follow-up.)
Completed | 0 | 0
Not Completed | 107 | 114
Not completed — Incomplete due to study termination | 107 | 114

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement | Total
Number analyzed (Participants) | 202 | 200 | 402
Age, Continuous [Mean (Full Range); unit: years] | 73 [46 to 93] | 76 [54 to 95] | 75 [46 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 142 | 269
  Male | 75 | 58 | 133

OUTCOME MEASURES:

1. Secondary Outcome: Harris Hip Score Pain
Description: Harris Hip Score Pain is detailed below as mean score for the Harris Hip Score Pain question. 44 being the highest score, and 0 being the lowest score. 44 is considered "None/Ignores." 40 is considered "Slight/Occasional." 30 is considered "Mild." 20 is considered "Moderate." 10 is considered "Marked." 0 is considered "Totally Disabled."
Time Frame: Pre-Operative, 6 months, 1 year, 2 year, 4 year, 6 year, 8 year, 10 year
Population: This population represents patients that returned for follow-up per protocol.
Measure: Mean (Standard Deviation); unit: Mean Hip Pain
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Number analyzed (Participants) | 202 | 200
Mean Hip Pain
  Pre-Operative Harris Hip Score Pain | 15.89 (7.64) | 14.74 (7.78)
  6 Month Harris Hip Score Pain | 39.78 (4.06) | 36.25 (9.69)
  1 Year Harris Hip Score Pain | 37.89 (9.54) | 37.76 (9.24)
  2 Year Harris Hip Score Pain | 36.93 (9.47) | 34.59 (10.54)
  4 Year Harris Hip Score Pain | 38.38 (9.78) | 41.27 (4.22)
  6 Year Harris Hip Score Pain | 44.00 (0) | 42.00 (2.83)
  8 Year Harris Hip Score Pain | 37.00 (9.90) | NA (NA) — No patients were analyzed at this time interval

2. Primary Outcome: Harris Hip Score
Description: The Harris Hip Score is detailed below as a range. 100 being the highest score, and 0 being the lowest score. 90-100 is considered "Excellent." 80-89 is considered "Good." 70-79 is considered "Fair." Less than 70 is considered "Poor."
Time Frame: 10 Years Post-Operative
Population: This population represents patients that returned for follow-up per protocol. Because no patients returned at the primary outcome measure time frame (10 years), 0 patients were analyzed at 10 years.
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 Years
Arm/Group | Answer Stem Utilizing Simplex Cement | Answer Stem Utilizing Palacos Cement
Serious Adverse Events (participants affected / at risk) | 15/202 | 8/200
Other Adverse Events (participants affected / at risk) | 0/202 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Answer Stem Utilizing Simplex Cement (N=202) | Answer Stem Utilizing Palacos Cement (N=200)
Dislocation (Musculoskeletal and connective tissue disorders) | 9 (31) | 1 (1)
Femoral loosening (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Deep infection < 6 weeks (Infections and infestations) | 1 (1) | 2 (2)
Deep infection > 6 weeks (Infections and infestations) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Femoral, acetabular loosening and instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Revision with all components removed and re-implantation (Surgical and medical procedures) | 0 (0) | 2 (2)
I&D, exchange of poly liner (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated prematurely after sponsor no longer distributed the products involved and follow-up failed to produce sufficient data to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can conduct a pre-publication review of articles, papers, or presentations which the PI desires to publish. Any such review must be completed by sponsor within thirty (30)days of the submission of the request. The PI must include whatever credits the sponsor deems necessary or appropriate to disclose its proprietary interest to the material disclosed in the article, paper or presentation.